CLINICAL TRIAL: NCT05580991
Title: A Phase 1, Dose Escalation, Open-Label Study of Intratumoral CAN1012 in Subjects with Unresectable or Metastatic Advanced Solid Tumors
Brief Title: Intratumoral CAN1012(selective TLR7 Agonist) in Subjects with Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Canwell Biotech Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KW-CAN1012-101
Record Dates: First submitted 2022-10-10; First posted 2022-10-14 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- CAN1012 (Experimental): CAN1012 intratumoral injection given alone
  Interventions: Drug: CAN1012

INTERVENTIONS:
Drug: CAN1012 — CAN1012 IT injection (once every 4 weeks)

SUMMARY:
To evaluate CAN1012 when administered by IT injection to subjects with advanced solid tumors who are not candidates for standard therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female age >18 years at screening.
2. Metastatic or locally advanced solid tumor that has progressed on, is refractory to, or for which there is no efficacious standard of care therapy.
3. At least one measurable lesion (RECIST 1.1)
4. At least one lesion that can receive intratumor injection multiple times
5. Performance status of 0 or 1 on the ECOG Performance Scale.
6. Life expectancy >12 weeks at Baseline.
7. Demonstrate adequate organ function as defined below. All screening laboratory assessments should be performed within 14 days of treatment initiation and include the following:

   1. Absolute neutrophil count (ANC) >=1.5 × 10^9/L； Platelets >=100 × 10^9/L；Hemoglobin >=9 g/dL;
   2. Measured or calculated creatinine clearance (CrCl) >=60 mL/min;
   3. Total bilirubin ≤1.5 × ULN OR direct bilirubin ≤ULN for subjects with total bilirubin levels > 1.5× ULN； Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 × ULN OR ≤5 × ULN for subjects with liver metastases."
8. Women of childbearing potential must have negative serum pregnancy test within 3 days prior to receiving the first study drug administration.For women of childbearing potential, must be willing to use an adequate method of contraception from 30 days prior to the first study drug administration and 120 days following last day of study drug administration.Male subjects of childbearing potential must be surgically sterile or must agree to use adequate method of contraception during the study and at least 120 days following the last day of study drug administration.
9. Able and willing to provide written informed consent and willing to comply with the study's requirements.

Exclusion Criteria:

1. Have a history of allergies in the past, and known to be allergic to CAN1012 injection or any of its components.
2. Have received TLR7/8 agonists in the past (except for topical dermal medications).
3. A history of another malignancy within the past 3 years that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin that has undergone curative therapy, or in situ cervical cancer.

"4. Unstable/inadequate cardiac function defined as follows:

1. New York Heart Association Class 3 or 4 congestive heart failure
2. uncontrolled hypertension
3. acute coronary syndrome within 6 months
4. clinical important cardiac arrhythmia
5. mean corrected QT (QTc) interval corrected for heart rate > 450 msec (m) or > 470 msec (md)." 5. Has known active infection with the human immunodeficiency virus, Hepatitis B(e.g., hepatitis B surface antigen [HBsAg] reactive) or Hepatitis C (e.g., hepatitis C virus [HCV] ribonucleic acid [qualitative] is detected), or active coronavirus disease 2019(COVID-19) infection. Note: Subjects who have been vaccinated against Hepatitis B and who are positive only for the Hepatitis B surface antibody are permitted to participate inthe study.

   6. Participated in a clinical study of an investigational agent within 4 weeks of screening.

   7. Have received chemotherapy, radiotherapy, biological therapy, endocrine therapy, targeted therapy, immunotherapy and other anti-tumor therapy within 4 weeks before the first administration of the research drug [among them, the following provisions are: nitrosourea (such as carmustine, lomustine, etc.) or mitomycin C is within 6 weeks before the first administration of the research drug; Oral fluorouracil, small molecule targeted drugs are 5 half-lives (whichever is longer) for 2 weeks before the first administration of the study drug or the known drug; Traditional Chinese medicines with antitumor indications are within 2 weeks before the first administration of the study drug].

   8. Has an active infection requiring systemic therapy within 4 weeks before the first dose of the drug under study, including but not limited to complications of infection that require hospitalization, bacteremia, severe pneumonia, etc.

   9. Patients with symptoms or who have undergone radiation therapy or surgery within 3 months prior to the first administration of the study (those with brain metastases and instability shall not be included).

   10. Injections of primary or metastatic lesions should be avoided in the central nervous system, thoracic cavity, heart and large blood vessels, liver, lungs, spleen and pancreas.

   11. Unresolved toxicities from prior therapy, defined as having not resolved to Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0 (v5.0) Grade 0 or 1, with exception of endocrinopathies from prior therapy, alopecia, and vitiligo.

   12. Treatment with systemic corticosteroids at doses exceeding 10 mg/day prednisone or equivalent.

   13. Uncontrolled concurrent illness 14. Patients with clinically significant lung diseases in the past, including but not limited to interstitial lung disease, pulmonary fibrosis and severe radiation pneumonitis.

   15. A history of coagulopathy resulting in uncontrolled bleeding or other bleeding disorders.

   16. Concomitant or planned use of sensitive substrates of major cytochrome P450 enzymes (see Appendix 4).

   17. Has known psychiatric, substance abuse, or other disorders that would interfere with cooperation with the requirements of the study in the opinion of the investigator.

   18. Persons with a known history of alcohol or drug dependence. 19. Is pregnant or breastfeeding. 20. The investigator believes that the subject is unsuitable for other reasons to participate in this clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2022-09-09 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Safety as determined by assessment of dose limiting toxicities per protocol of CAN1012 with cancers. | 12 months
  Safety as determined by assessment of dose limiting toxicities per protocol of CAN1012 with cancers.
Tolerability as determined by assessment of the maximum tolerated dose or maximal assessed dose per protocol of CAN 1012 with cancers. | 12 months
  Tolerability as determined by assessment of the maximum tolerated dose or maximal assessed dose per protocol of CAN 1012 with cancers.
Recommended Phase 2 Dose (RP2D) | 12 months
  To determine a recommended phase 2 dose of CAN1012 for further development by evaluating number of patients with treatment-related adverse events as assessed by the Common Terminology Criteria for Adverse Events version 5.0 (CTCAE 5.0)
Maximum Tolerated Dose (MTD) | 12 months
  Determine the maximum tolerated dose by assessing the Incidence of Dose Limiting Toxicities (DLTs), treatment emergent and treatment related adverse events (assessed by CTCAE 5.0).
PK characterization - Cmax | 12 months
  Maximum observed plasma and tumor concentration of CAN1012 after IT administration.
PK characterization - tmax | 12 months
  Time to reach maximum plasma and tumor concentration of CAN1012 after IT administration.
tumor size in injected lesions and non-injected lesions | 12 months
  Changes in tumor size using computed tomography (CT) scan or magnetic resonance imaging (MRI) scan assessment based on Response Evaluation Criteria in Solid Tumors (RECIST) v1.1

CONTACTS AND LOCATIONS:
Locations (1):
- Canwell Biotech Limited, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No